CLINICAL TRIAL: NCT04266509
Title: PHASE 1, OPEN-LABEL, FIXED-SEQUENCE STUDY TO EVALUATE THE EFFECT OF REPEAT-DOSE RIFAMPIN ON THE PHARMACOKINETICS OF PF-06651600 IN HEALTHY PARTICIPANTS
Brief Title: Study to Evaluate the Effect of Repeat-Dose Rifampin on the Pharmacokinetics (PK) of PF-06651600
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: B7981026; 2019-004643-72 (EudraCT Number)
Record Dates: First submitted 2020-02-10; First posted 2020-02-12 (Actual); Last update posted 2020-09-16 (Actual); Status verified 2020-09

CONDITIONS: Healthy Volunteers
Keywords: PF-06651600; Rifampin; Drug-drug interaction study; Pharmacokinetics
MeSH Terms: interventions — PF-06651600; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Rifampin and PF-06651600 DDI (Experimental): In Period 1, participants will receive a single oral 50 mg dose of PF-06651600. In Period 2, participants will receive rifampin 600 mg QD in the mornings of Day 1 to Day 7, in the morning of Day 8 participants will be administered with rifampin 600 mg 2 hour prior to administration of a single 50 mg oral dose of PF-06651600.
  Interventions: Drug: PF-06651600; Drug: Rifampin

INTERVENTIONS:
Drug: PF-06651600 — 50 milligram (mg) tablet
Drug: Rifampin — 600 mg provided as two 300 mg capsules.
  Other Names: Rifadin®.

SUMMARY:
Study to Evaluate the Effect of Repeat-Dose Rifampin on the pharmacokinetics (PK) of PF-06651600.

ELIGIBILITY:
Inclusion Criteria:

* Male and/or female participants who are healthy as determined by medical evaluation including medical history, full physical examination which includes BP and pulse rate measurements, clinical laboratory tests, and 12-lead ECG.
* BMI of 17.5 to 30.5 kg/m2; and a total body weight >50 kg (110 lb).

Exclusion Criteria:

* Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurological, dermatological or allergic disease (including drug allergies, but excluding untreated, asymptomatic, seasonal allergies at the time of dosing).
* Any condition possibly affecting drug absorption (eg, gastrectomy, cholecystectomy).
* Systemic therapy with any of the medications that are moderate or strong CYP3A4 and/or CYP2C19 inhibitors within 28 days or 5 half-lives (whichever is longer) or moderate or strong CYP3A and/or CYP2C19 inducers within 28 days or 5 half-lives (whichever is longer) prior to the first dose of investigational product.
* Known participation in a clinical trial of PF-06651600 within 60 days prior to the first dose of investigational product; participation in any clinical trail of PF-06651600 and the participant experienced AE that led to discontinuation, or had SAE, that in the judgment of the investigator were PF-06651600-related.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2020-06-25 (Actual); Primary Completion 2020-09-10 (Actual); Study Completion 2020-09-10 (Actual)

PRIMARY OUTCOMES:
Cmax (maximum plasma concentration) of PF-06651600 | Hour 0, and 0.25, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours post post Period 1, Day 1, Period 2, Day 8.
AUC (Area under the curve) of PF-06651600 | Hour 0, and 0.25, 0.5, 1, 2, 3, 4, 5, 6, 8, 10, 12, 24 hours post post Period 1, Day 1, Period 2, Day 8.
  Area under the plasma concentration-time profile from time 0 extrapolated to infinite time.

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Brussels Clinical Research Unit, Brussels, Bruxelles-capitale, Région de, Belgium

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B7981026